CLINICAL TRIAL: NCT07316374
Title: Evaluation of AI-Based Chatbots for Improving Anxiety-Related Mental Health Literacy: A Randomized Controlled Trial
Brief Title: AI Chatbots for Anxiety Mental Health Literacy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Anxiety Literacy AI Chatbot
Record Dates: First submitted 2025-12-16; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Anxiety Literacy; Anxiety Disorders; Mental Health Literacy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AI Educator Only (Experimental): Participants will interact with the AI-powered psychoeducation chatbot for one week. The chatbot delivers structured conversational modules covering anxiety concepts, symptoms, causes, treatment options, and self-help strategies.
  Interventions: Behavioral: AI Anxiety Literacy Education
- AI Educator + AI Anxiety Friend Simulators (Experimental): Participants will first complete all AI Educator modules and then interact with five AI Anxiety Friend Simulators over one week. Each simulator represents a distinct anxiety presentation and prompts participants to identify symptoms, explore mechanisms, and propose support strategies.
  Interventions: Behavioral: AI Anxiety Literacy Education; Behavioral: AI Anxiety Friend Simulation
- Text-Based Psychoeducation (Active Comparator): Participants will receive standard text-based psychoeducation materials about anxiety, including definitions, symptoms, causes, and coping strategies, to be completed within one week.
  Interventions: Behavioral: Text-Based Anxiety Psychoeducation

INTERVENTIONS:
Behavioral: AI Anxiety Literacy Education — AI Anxiety Literacy Education is an AI-powered, psychologically informed chatbot designed to improve mental health literacy related to anxiety through conversational education.
  The chatbot delivers structured modules covering the definition of anxiety, common cognitive, emotional, physical, and behavioral symptoms, contributing factors, treatment options, and practical self-help strategies.
  Content is presented in non-clinical language and adapted to user responses through guided questions and feedback, encouraging users to reflect on their own experiences.
  Arms: AI Educator + AI Anxiety Friend Simulators; AI Educator Only
Behavioral: AI Anxiety Friend Simulation — AI Anxiety Friend Simulation is an AI-powered conversational intervention designed to allow participants to practice recognizing and responding to anxiety-related experiences in a simulated interaction. The chatbot role-plays individuals experiencing different anxiety presentations and communicates in a natural, everyday manner that may include uncertainty, emotional reactions, or defensiveness.
  Participants are guided to identify anxiety symptoms, explore causes, and propose supportive responses. The chatbot provides feedback and prompts reflection based on participants' responses. Participants access the simulation online and complete multiple simulated conversations over a one-week period.
  Arms: AI Educator + AI Anxiety Friend Simulators
Behavioral: Text-Based Anxiety Psychoeducation — Text-Based Anxiety Psychoeducation consists of written educational materials providing information about anxiety in a non-clinical, accessible format. The materials cover the definition of anxiety, common cognitive, emotional, physical, and behavioral symptoms, contributing factors, and general coping and self-help strategies. Participants access the materials online and are instructed to review all content within a one-week period. The materials are static and do not provide interactive feedback or personalized responses.
  Arms: Text-Based Psychoeducation

SUMMARY:
The goal of this clinical trial is to examine whether AI-based chatbots can improve anxiety-related mental health literacy in adults with varying levels of anxiety. The study aims to learn whether interactive AI chatbots can improve understanding of anxiety, attitudes toward anxiety, help-seeking intentions, confidence in supporting others, and anxiety symptoms, compared with standard text-based educational materials.

The main questions it aims to answer are:

1. Does an AI-based psychoeducation chatbot improve anxiety-related mental health literacy compared with text-based psychoeducation?
2. Does adding interactive anxiety simulation conversations further improve mental health literacy and related outcomes compared with psychoeducation alone?

Researchers will compare participants who use an AI psychoeducation chatbot alone, participants who use an AI psychoeducation chatbot combined with anxiety simulation chatbots, and participants who receive text-based psychoeducation, to see whether the AI-based interventions lead to greater improvements in mental health literacy and related outcomes.

Participants will:

1. Complete baseline questionnaires assessing anxiety-related knowledge, attitudes, and symptoms
2. Be randomly assigned to one of three groups: AI psychoeducation chatbot, AI psychoeducation chatbot plus anxiety simulation chatbots, or text-based psychoeducation
3. Use the assigned intervention over a one-week period
4. Complete follow-up questionnaires immediately after the intervention and at later follow-up time points

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years.
2. Able to use digital devices (e.g., smartphone or computer) to complete AI-based conversations and questionnaires.
3. Willing to participate in a one-week online intervention.
4. Proficient in Chinese and able to understand study instructions and provide informed consent.
5. Participants with varying levels of anxiety symptoms are eligible.

Exclusion Criteria:

1. Self-reported history of severe psychiatric disorders (e.g., psychotic disorders, bipolar disorder).
2. Currently receiving psychological or psychiatric treatment.
3. Severe mental health symptoms requiring immediate clinical intervention.
4. Inability to use mobile or internet-enabled devices independently.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety Literacy Scale (ALS) | pre-intervention, post-intervention (1-week), 4-week follow-up, 12-week follow-up
  The Anxiety Literacy Scale is a 22-item questionnaire designed to assess individuals' knowledge about anxiety. Each statement is answered using a binary response format (true or false). For each item, participants are also asked to rate their certainty in their response on a 5-point Likert scale. Correct responses are summed to produce a total knowledge score, with higher scores indicating greater anxiety-related mental health literacy. Certainty ratings are used to assess participants' confidence in their knowledge and to examine the calibration between knowledge accuracy and subjective certainty.
Anxiety Stigma Scale | pre-intervention, post-intervention (1-week), 4-week follow-up, 12-week follow-up
  The Anxiety Stigma Scale is designed to measure stigma associated with Anxiety. It has two subscales which measure two different types of stigma: personal and perceived. The Personal Stigma Subscale measures stigma in the respondents own attitudes towards anxiety by asking them to indicate how strongly they personally agree with ten statements about anxiety.
  The Perceived Stigma Subscale measures the respondent's perception about the attitudes of others towards anxiety by asking them to indicate what they think most other people believe about the same ten statements.
  Responses to each item are measured on a five-point scale (ranging from zero 'strongly disagree' to four 'strongly agree'). Higher scores indicate higher levels of depression stigma.
Adapted General Help-Seeking Questionnaire | pre-intervention, post-intervention (1-week), 4-week follow-up, 12-week follow-up
  The General Help-Seeking Questionnaire (GHSQ) in this study is an adapted 17-item version designed to fit Chinese cultural contexts. It assesses an individual's intentions to seek help for personal or emotional problems from both formal sources (e.g., mental health professionals, doctors) and informal sources (e.g., family, friends). Each item is rated on a 7-point Likert scale, ranging from 1 ("Extremely Unlikely") to 7 ("Extremely Likely"), with higher scores indicating a greater likelihood of seeking help.
Confidence in Helping Others | pre-intervention, post-intervention (1-week), 4-week follow-up, 12-week follow-up
  The Confidence in Helping Others Scale is a self-developed, 13-item questionnaire designed to measure participants' confidence in providing support to individuals experiencing mental health issues. Each item is rated on a 5-point Likert scale, ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"), with higher scores indicating greater confidence in recognizing symptoms, offering emotional support, and encouraging help-seeking.
Mental Health Self-efficacy Scale | pre-intervention, post-intervention (1-week), 4-week follow-up, 12-week follow-up
  The Mental Health Self-efficacy Scale is a 6-item questionnaire designed to measure participants' confidence in effectively manage stress, anxiety or depression about themself. Each item is rated on a 10-point Likert scale, ranging from 1 ("Not at all confident") to 10 ("Totally confident"), with higher scores indicating greater confidence in self-efficacy about mental health.
Bot Usability Scale | post-intervention (1-week)
  The Bot Usability Scale (BUS) in this study is an adapted 11-item version designed to assess the usability of AI-based chatbots. It evaluates participants' perceptions of the ease of use, effectiveness, efficiency, and overall user experience of the chatbots. The scale uses a 5-point Likert scale, ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"), with higher scores indicating better perceived usability. Participants will complete the adapted BUS separately for both the AI Educator and the AI Anxiety Friend Simulators. The adapted BUS maintains the core usability assessment principles of the original scale while being tailored for AI-driven conversational agents.

SECONDARY OUTCOMES:
General Anxiety Disorder (GAD-7) | pre-intervention, post-intervention (1-week), 4-week follow-up, 12-week follow-up
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report questionnaire used to assess the severity of generalized anxiety symptoms over the past two weeks. Each item corresponds to common symptoms of generalized anxiety disorder (GAD) and is rated on a 4-point Likert scale, ranging from 0 ("Not at all") to 3 ("Nearly every day"), with higher scores indicating greater symptom severity.
Patient Health Questionnaire (PHQ-9) | pre-intervention, post-intervention (1-week), 4-week follow-up, 12-week follow-up
  The Patient Health Questionnaire (PHQ-9) consists of 9 items designed to assess the severity of depressive symptoms over the past two weeks. Each item corresponds to one of the nine DSM-5 criteria for major depressive disorder and is rated on a 4-point Likert scale, ranging from 0 ("Not at all") to 3 ("Nearly every day"), with higher scores indicating greater symptom severity.
Intolerance of Uncertainty Scale | pre-intervention, post-intervention (1-week), 4-week follow-up, 12-week follow-up
  Intolerance of Uncertainty Scale is designed to measure participants' attidudes about uncertaunty. It is a self-developed, 12-item questionnaire, ranging from 1 ("not at all characteristic for me")) to 5 ("entirely characteristic of me"), with higher scores indicating greater intolerance.
Negative Effects Scale, NES | post-intervention (1-week)
  Sometimes programs that aim to improve mental health can also have unwanted effects.The Negative Effects Scale (NES) is a 6-item self-report assessment tool designed to measure the participants' perceptions of unwanted experience. Each item is rated on a 5-point Likert scale, ranging from 1 (" Not at al") to 5 ("Extremely severe"), with higher scores indicating a greater negative Effects.
Basic Empathy Scale in Adults (BES-A) | pre-intervention, post-intervention (1-week), 4-week follow-up, 12-week follow-up
  The Basic Empathy Scale in Adults (BES-A) is a 20-item self-report questionnaire designed to assess an individual's capacity for empathy, including both cognitive empathy (understanding others' emotions) and affective empathy (sharing others' emotions). Each item is rated on a 5-point Likert scale, ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"), with higher scores indicating greater empathy.
Mental Health Behavior | pre-intervention, 4-week follow-up, 12-week follow-up
  This questionnaire is self-conducted and assesses the frequency of various mental health-related behaviors over the past month. Participants rate each behavior based on how often they engaged in it, using a 5-point scale (0 = Never, 4 = More than 4 times per week). The results provide insight into individuals' proactive engagement in mental well-being practices.

OTHER OUTCOMES:
Peking alexithymia scale | pre-intervention
  The Peking Alexithymia Scale (PAS) is a culturally adapted assessment tool designed to measure alexithymia-a personality construct characterized by difficulties in identifying and describing one's own emotions, coupled with an externally oriented thinking style-among Chinese populations. This subscale consists of 9 items divided into three distinct dimensions, each targeting a core feature of alexithymia.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university, Beijing, China

IPD SHARING:
Plan to Share IPD: No